CLINICAL TRIAL: NCT03121521
Title: The Effects of Melatonin on Elevated Liver Enzymes During Statins Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Cezary Chojnacki, Head of Department of Clinical Nutrition and Gastroenterological Diagnostics, Medical University of Lodz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN 402 54 37/40; RNN/45/12/KB (Other: Bioethics Committee of the Medical University in Lodz)
Record Dates: First submitted 2017-04-13; First posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Hepatopathy
Keywords: statins liver enzymes melatonin
MeSH Terms: conditions — Digestive System Diseases | interventions — Melatonin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- melatonin (Experimental): Melatonin 10mg/d p.o.
  Interventions: Drug: Melatonin 10 mg
- placebo (Placebo Comparator): placebo 10mg/d p.o.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin 10 mg — melatonin 10mg daily p.o.
  Other Names: Melatonin Lek-AM 10mg
  Arms: melatonin
Drug: Placebo — Placebo 10mg daily p.o.
  Other Names: Placebo 10mg
  Arms: placebo

SUMMARY:
Introduction. Statins are generally well tolerated but not devoid of side effects. Quite often it is manifested by asymptomatic increase in the level of aspartate and alanine aminotransferase. In such cases patients to administer hepatoprotective drugs, but most of them used for this purpose are ineffective. The aim of this study was assess the usefulness of melatonin in counteracting the adverse hepatic events from statins. Methods. The research program included 60 patients(aged 47-65 years, 41 women and 23 men)with hyperlipidemia taking atorvastatin or rosuvastatin in dose 20-40 mg daily. The patients were randomly allocated in two groups. Group I (n=30) was recommended to take the same statin at a standardized daily dose of 20 mg together with melatonin at a dose 2 x 5 mg, at 7:00 and 21:00. In group II (n=30) patients took statins with placebo at the same time of the day. Follow-up laboratory tests (AST, ALT, GGT, ALP, cholesterol, triglycerides) were evaluated after 2,4 and 6 mounts of treatment.

DETAILED DESCRIPTION:
Introduction Statins are widely used in the treatment and prevention of lipid metabolism disorders. They are generally well tolerated but not devoid of side effects. These include, among others, muscular symptoms, arthritis, headaches, gynecomastia. Myositis and rhabdomyolysis associated with increased activity of creatinine kinase and serum creatinine levels are rare but serious adverse events of statin therapy. The risk of these complications is increased in elderly patients with chronic diseases and in alcohol abusers.

Furthermore, statins cause hepatotoxic effect which is observed in several percent of treated patients, usually in the first weeks of the therapy . Most frequently it is manifested by asymptomatic increase in the level of aspartate and alanine aminotransferase. This is usually a temporary increase, but in some patients the level of these enzymes exceeds 3 times the normal limit, which is a matter of concern. In such cases, patients expect the decision to discontinue the treatment or to administer hepatoprotective drugs. Acetylcholine, sylibinin, phospholipids and other drugs used for this purpose are not always effective. Therefore, there is still search for alternative drugs for the protection of liver.

In own study melatonin was used for this purpose because previous experimental studies had demonstrated that it protected liver against harmful effects of many toxic agents as well as the consequences of ischemia-reperfusion model.

The liver is an organ in which there comes to intensive metabolic and detoxification processes. In their course large amounts of reactive oxygen species are generated and they exert a toxic effect on hepatocytes. A complex antioxidant system - in which metabolized there melatonin (pineal and from other sources) is an important part - prevents that.

The main melatonin metabolic pathway in the liver is through hydroxylation pathway at the C-6 position by 6-hydroxylase and P450 cytochromes (CYP1A1, CYP1A2, CYP2P19, CYP1B1 isozymes). The 6-hydroxymelatonin, formed in this process, is conjugated with sulphate and glucuronide to 6-hydroxymelatonin sulphate or glucuronide. In this process melatonin and its metabolites exert high antioxidant activity.

An alternative metabolic pathway includes melatonin oxidation to N-acetyl-formyl-5- methoxykynuramine (AFMK) and N-acetyl-5-methoxykynuramine (AMK). The kynurenine pathway of melatonin metabolism leads to formation of a series of free radical scavengers.

Furthermore, melatonin decreases the production of proinflammatory cytokines and inhibits hepatic fibrogenesis. Owing to its multidirectional action in liver, apoptosis and necrosis decrease, the integrity is protected and regeneration is improved.

The aim of this study was to assess the usefulness of melatonin in counteracting the adverse hepatic events from statins.

Material and Methods Patients and Data Collection The research program included 30 subjects, aged 47-68 years, 41 women and 23 men. All women were I the postpostmenopausal period. Recruitment and diagnostic tests were conducted in the Department of Gastroenterology, Medical University of Lodz and Outpatient Consulting Clinic "Gastro" in Lodz.

The research study was performed in the years 2012-2016. Therapeutic Procedures After inclusion into the study, all patients were recommended the same balanced diet with limited animal fats and simple carbohydrates of caloric content of 1600 kcal. At the same time, they were recommended to continue the treatment with the same statin at a daily dose of 20 mg.

The patients were randomly allocated into two groups. Group I (n=30) was recommended to take statin together with melatonin (LEK-AM, Poland) at a dose of 2x5 mg, at 7:00 a.m. and 9:00 p.m. In Group II (n=30) patients took statin with placebo (LEK-AM, Poland) at the same dose and time of the day.

Follow-up laboratory tests (AST, ALT, GGT, ALP, cholesterol and triglycerides) were evaluated after 2,4 and 6 months of treatment.

Ethical procedures A written consent was obtained from the patients and the Bioethics Committee of the Medical University in Lodz approved the study protocol (RNN/45/12/KB).

Tests were conducted in accordance with the Declaration of Helsinki and with the principles of Good Clinical Practice.

Statistical analysis All parameters were checked for normality using the Shapiro-Wilk test. Wilcoxon's rank sum test was used for the comparison of basal treatment differences between each liver enzyme level. Comparison of parameters in four time series was calculated using ANOVA Friedman test. Mann-Whitney U test was used for nonparametric data to perform the comparison between groups. Calculation were made using Statistical 9.1 Microsoft Co. software, and statistical significance was established at p< 0,05.

Acknowledgments This work was supported by the grant from the Polish Ministry of Science and Higher Education No: NN 402 54 37/40.

Competing Interests The authors declare that they have no competing interests.

ELIGIBILITY:
Inclusion Criteria:- hyperlipidemia treated with statins for minimum 6 months

* at least 2-fold increase in the level of aspartate and alanine aminotransferase found in two consecutive tests
* the persistence of increased aminotransferase levels despite the reduction in the statin dose At the time of the inclusion of patients in the study, 38 subjects were taking atorvastatin ( 20 mg), and 26 - rosuvastatin at the dose 40 mg (3 patients), - 20mg (19 patients) and 15 mg (4 patients).

Exclusion Criteria:- history of viral hepatitis

* cholelithiasis 4
* body mass index (BMI)>30kg/m2
* alcohol abuse
* familial hypercholesterolemia
* established hypertension
* thyroid diseases
* other organic, metabolic or mental diseases
* hormone replacement therapy
* taking other medications, especially analgesics and psychotropic drugs

Ages: 47 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
liver enzymes | 6 months
  levels